CLINICAL TRIAL: NCT05646498
Title: Clinical and Patient- Satisfaction Outcomes During Management of Atrophied Unilateral Distally Extension Maxillary Ridge With Two Different Minimal Invasive Treatment Modalities. 1-year Randomized Controlled Clinical Trial.
Brief Title: Management of Distally Extension Maxillary Atrophied Ridge With Two Different Minimal Invasive Treatment Modalities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elgamal, Associate professor of removable prosthodontics, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A01140420
Record Dates: First submitted 2022-11-17; First posted 2022-12-12 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Partial Edentulism Class 2 Due to Periodontal Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implant retained removable overdentures (Active Comparator): Procedure: Long implant and partial overdentures insertion of long implants anterior to the maxillary sinus to retain partial overdentures
  Device: Partial overdentures Distal extension metallic partial dentures retained by attachments to the implants
  Interventions: Procedure: Closed sinus lift procedure; Device: Crestal sinus lift
- implant supported fixed screw retained prosthesis (Active Comparator): Procedure: Sinus lift and long implant performing sinus lift surgical procedure with simultaneous placement of limplants to support screw-retained prosthesis
  Device: Metal ceramic prosthesis on long implants porcelain fused to metal fixed screw-retained prosthesis supported by implants
  Interventions: Procedure: Closed sinus lift procedure; Device: Crestal sinus lift

INTERVENTIONS:
Procedure: Closed sinus lift procedure — The closed sinus lift is the elevation of the sinus membrane through the osteotomy
  Other Names: Minimal invasive sinus lift
Device: Crestal sinus lift — The crestal approach is the elevation of the sinus membrane by osteotomes, piezosurgery, or Densah burs.
  Other Names: Minimal invasive sinus lift

SUMMARY:
This study will compare clinical and radio graphic outcomes of two minimally invasive different treatment modalities for atrophied unilateral distal extension maxillary ridges these modalities include

1. Medially placed implant and Implant retained distal extension removable partial denture
2. Sinus lift and long implant to support fixed screw-retained prosthesis

DETAILED DESCRIPTION:
Patient selection:

For this study, 40 patients were selected from the clinic of Prosthodontics Department, Faculty of Dentistry, Mansoura University.

Inclusion criteria:

The patients will be selected according to the following:

* They have atrophied unilateral distal extension maxillary ridge and remaining alveolar bone height 6- 8 mm as verified by preoperative cone beam. They are healthy, free from any systemic diseases relating to the bone resorption (diabetes - hyperparathyroidism). This can be achieved through medical history and clinical examination by a physician and laboratory investigations.
* Posterior maxillary alveolar ridge deficient in height, width and covered with healthy firm covering.
* Patients are less satisfied with conventional removable partial denture.
* Absence of maxillary sinus diseases. Exclusion criteria

Patients were not eligible for this work if any of the following criteria were met:

* Acute or chronic sinus pathology
* History of a sinus augmentation in the past in the relevant sinus
* Poor dental hygiene. Smoker.
* Compromised general health (uncontrolled diabetes, bleeding disorder….). All patient were informed about all procedures that will be done and they sign the written consent form of ethical committee in faculty of dentistry Mansoura university.

Three treatment groups will be classified randomly, as follow:

* Group I: patients received one implant in premolar area medial to maxillary sinus and used to retain partial over-denture.
* Group II: patient underwent sinus lift and receive screw retained prosthesis on long implant All implants were inserted using computer guided and flap-less implant surgery and conventional loading protocol was used.

Evaluation methods Clinical and radio-graphic evaluation

1. Modified Plaque index. Assessment of plaque accumulation with a modified plaque index : Score 0: No detection of plaque, Score 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant, Score 2 Plaque can be seen by a naked eye, Score 3 Abundance of soft matter.
2. Marginal index. Assessment of bleeding tendency with a modified bleeding index : Score 0 No bleeding when a periodontal probe is passed along the margin adjacent to the implant. Score 1 Isolated bleeding spot visible, Score 2 Blood forms a confluent red line on margin, Score 3 Heavy or profuse bleeding.
3. Attachment level. Distance from the junction implant/crown to the most apically probe able portion, in millimeters.
4. Pocket depth. Distance between the margin and the most apically probable portion, in millimeters Assessed by insertion of a standard periodontal probe with a point diameter of 0.5 mm using a probing force of 0.5 N.
5. Implant stability quotient. Using resonance frequency analysis b- Radio-graphic evaluation will be performed in terms of:

Vertical bone loss will be evaluated as follows:

The distance between implant plate form and first bone to implant contact will be evaluated after one year.

ELIGIBILITY:
Inclusion Criteria:

* The patients will be selected according to the following:

  * They have atrophied unilateral distal extension maxillary ridge and remaining alveolar bone height 6- 8mm as verified by preoperative CBCT, They are healthy, free from any systemic diseases relating to the bone resorption (diabetes - hyperparathyroidism). This can be achieved through medical history and clinical examination by a physician and laboratory investigations.
  * Posterior maxillary alveolar ridge deficient in height, width and covered with healthy firm mucosa.
  * Patients are less satisfied with conventional RPD.
  * Absence of maxillary sinus diseases.

Exclusion Criteria:

* • Acute or chronic sinus pathology

  * History of a sinus augmentation in the past in the relevant sinus
  * Poor dental hygiene. Smoker.
  * Compromised general health (uncontrolled diabetes, bleeding disorder

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-06-22 (Estimated)

PRIMARY OUTCOMES:
Plaque index evaluation | one year
  measuring plaque accumulation around implants using scores Plaque will be assessed according to modified plaque index describe as follows: score 0; no plaque detected, score 1; plaque recognized only by running a probe across a smooth marginal surface of the implant, score 2; plaque can be seen by naked eye, and score 3; abundance of soft mater.
Gingival index evaluation | one year
  measuring inflammation around implants using scores Modified index will be recorded as follows: score 0; normal , score 1; mild inflammation (slight change in color & slight edema), but no bleeding on probing, score 2; moderate inflammation (redness & edema), and bleeding on probing, and score 3; sever inflammation (marked redness, edema & ulceration) with tendency to spontaneous bleeding.
Probing depth evaluation | one year
  measuring per-implant probing depth in mm. Using a calibrated plastic periodontal probe, the distance between marginal border of the and the tip of the probe was measured in mm and considered as pocket depth.
Implant stability evaluation | one year
  measuring the mobility of the implants using resonance frequency analysis Implant stability quotient) The resonance frequencies will be measured with the osstell® device (implant stability meter) and will be expressed with measurement scale (implant stability quotient).
Radio graphic evaluation | one year
  measuring bone loss around implants in mm Radio-graphs were taken using direct digital imaging system
  - Marginal alveolar bone changes (vertical and horizontal bone loss) were measured at medial and distal surface of each implant in mm.
Patient satisfaction | one year
  Patient satisfaction using questionnaire (visual analogue scale) Patient satisfaction was evaluated using a questionnaire based on visual analog scale . Patients were asked to mark their answer (amount of satisfaction) on a 100-mm line (with zero refers to not satisfied at all and 100 refers to completely satisfied). The mean of the answers (length of the lines from zero to the marks in mm) for each question. complete satisfaction). The questions cover several items related to prosthesis such as: retention, stability, comfort, ease of cleaning, ease of speaking, ease of chewing, limited activities due to embarrassment, quality of bolus and was subjected to statistical analysis

SECONDARY OUTCOMES:
Prosthetic complication | one year
  incidence of prosthetic aspects and maintenance requirements
Muscle activity | one year
  Muscle activity measure muscles activity in amplitude using electromyographs
maximum bite force | one year
  measuring maximum bite force in newton using bite force transducers

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University Mansoura, Eldakahlia, Egypt, 35516, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol